CLINICAL TRIAL: NCT07016919
Title: Early vs Conventional Enteral Nutrition After Uncomplicated Paediatric Open appendectomy-a Randomised Control Trial
Brief Title: Early vs Conventional Enteral Nutrition After Uncomplicated Paediatric Open Appendectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shaikh Zayed Hospital, Lahore (Other)
Responsible Party: Principal Investigator, Dr Noor Ulain, Doctor (Resident), Shaikh Zayed Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TERC/SC/INT/2025/360
Record Dates: First submitted 2025-06-01; First posted 2025-06-12 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Uncomplicated Acute Appendicitis in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Interventional group) early enteral nutrition (Experimental): Oral nutrition started within 6hours after surgery (paediatric open appendectomy) to this group
  Interventions: Other: early enteral nutrition
- Group B Conventional enteral nutrition (Active Comparator): Oral nutrition is started to this group after 24hours of the surgery (open appendectomy)
  Interventions: Other: Conventional enteral nutrition

INTERVENTIONS:
Other: early enteral nutrition — Oral nutrition started within 6hours after paediatric open appendectomy
  Arms: Group A (Interventional group) early enteral nutrition
Other: Conventional enteral nutrition — Oral nutrition started within 24hours after paediatric open appendectomy
  Arms: Group B Conventional enteral nutrition

SUMMARY:
This clinical trial is conducted to see if after surgery of appendix(open appendectomy) in children giving oral nutrition within 6hours of surgery instead of older method of starting oral nutrition after 24hours of surgery improves the outcome or not which is the length of hospital stay(from the day of surgery until discharge) and to look for complications associated with oral nutrition (nausea, vomiting, abdominal distension, diarrhea) as well as return of bowel activity after surgery that is passage of flatus(gas) and stool.Participants after taking informed consent are enrolled in two groups,group A in which oral nutrition is started in 6hours and group B in which oral nutrition is started after 24hours of surgery and then see for the outcome during hospital stay until 1week after discharge on follow up.

DETAILED DESCRIPTION:
All patients presenting to the department of paediatric surgery sheikh Zayed hospital with diagnosis of acute appendicitis fulfilling the inclusion criteria will be enrolled. Informed written consent will be taken from the patient's guardian or parent. Patients will be divided into two groups: group A Interventional group (early enteral nutrition) and group B control group (Conventional enteral nutrition). Both groups would be kept nothing per oral as per management of acute appendicitis. Pre-op antibiotic (injection ceftriaxone 50mg/kg/day) would be given. Patient would be kept pain free by using non opioid analgesics. Open appendectomy will be performed. The patients in group A will be given early enteral nutrition within 6hours after recovery from anesthesia and the patients in group B will be managed according to conventional perioperative management protocol of starting enteral nutrition 24hours post surgery. Data will be collected by the researcher along with the recording of results.Quantitative variables of the study would be length of hospital stay,time for the passage of stool and flatus after surgery and qualitative variables would be nausea, vomiting, diarrhea, abdominal distension,nasogatric tube insertion and readmission to hospital within 1week. All information will be collected through predesigned questionnaire. Data will be analyzed using Statistical Package for social sciences (IBM SPSS Statistics for windows,version 26.0).Data for age, hospital stay,time for the passage of flatus and stool will be described using mean±SD if normally distributed and median(IQR) otherwise.Comparison between groups will be made by using independent sample T-test or MannWhitney U test depending on normality of data. Data for qualitative measures like gender,nausea, vomiting, diarrhea, abdominal distension,NG tube insertion and readmission requirement will be described using frequency and percentages. Comparison among groups will be made by using Chi-square of Fisher-exact test depending on frequencies. P-value ≤ 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-14years
* Both male& female
* Uncomplicated appendicitis(no perforation/gangrene)
* patients who underwent open appendectomy
* ASA grade 1 only
* willing to participate and follow up

Exclusion Criteria:

* Any underlying comorbidities or organ dysfunction for example renal,GI, respiratory, congenital heart disease
* severe protein caloric malnourishment or obesity BMI>25
* any past surgical history related to gut
* any associated malignancy
* prolonged surgery(anesthesia time>3hours)
* complicated appendicitis (gangrene, perforation,intra-abdominal abscess)
* post-op shock
* ongoing infection
* GI dysfunction such as gastroesophageal reflux disease/obstruction.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | From enrollment until discharge from hospital (1-7days)
  Number of days from the day of surgery until the date of discharge (1-7days)

SECONDARY OUTCOMES:
Complications associated with early enteral nutrition | From enrollment until 1week after discharge on follow up
  Complications such as nausea, vomiting, abdominal distension and diarrhea associated with early enteral nutrition are observed
Time to return of bowel activity | From enrollment until discharge from hospital (1-7days)
  Time to return of bowel activity after surgery assessed by passage of flatus and stool

CONTACTS AND LOCATIONS:
Overall Officials: Dr Muhammad Ali sheikh, Study Director — Shaikh Zayed Hospital, Lahore
Locations (1):
- Shaikh Zayed federal postgraduate medical institute Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang SM, Chen J, Li H, Guo MF, Han N, Sun JS, Zhang CF, Su L. Clinical application of enhanced recovery after surgery concept in laparoscopic treatment of pediatric acute appendicitis. Pediatr Surg Int. 2023 Apr 11;39(1):178. doi: 10.1007/s00383-023-05439-5. PMID 37041392
- [Background] Mvoula L, Irizarry E. Tolerance to and Postoperative Outcomes With Early Oral Feeding Following Elective Bowel Surgery: A Systematic Review. Cureus. 2023 Aug 4;15(8):e42943. doi: 10.7759/cureus.42943. eCollection 2023 Aug. PMID 37667705
- [Background] Ying Y, Xu HZ, Han ML. Enhanced recovery after surgery strategy to shorten perioperative fasting in children undergoing non-gastrointestinal surgery: A prospective study. World J Clin Cases. 2022 Jun 6;10(16):5287-5296. doi: 10.12998/wjcc.v10.i16.5287. PMID 35812657
- [Background] Shang Q, Geng Q, Zhang X, Xu H, Guo C. The impact of early enteral nutrition on pediatric patients undergoing gastrointestinal anastomosis a propensity score matching analysis. Medicine (Baltimore). 2018 Mar;97(9):e0045. doi: 10.1097/MD.0000000000010045. PMID 29489656
- [Background] Lewis SJ, Egger M, Sylvester PA, Thomas S. Early enteral feeding versus "nil by mouth" after gastrointestinal surgery: systematic review and meta-analysis of controlled trials. BMJ. 2001 Oct 6;323(7316):773-6. doi: 10.1136/bmj.323.7316.773. PMID 11588077
- [Background] Mahmud GI, Hasan MM, Hakim MH, Rifat NH, Bhuiyan MAR, Islam T, Akter MN, Mithila SR, Mokarram MMB. The Outcome of Early Oral Feeding Following Elective Gastrointestinal Surgery. Cureus. 2024 Jul 4;16(7):e63802. doi: 10.7759/cureus.63802. eCollection 2024 Jul. PMID 39100012
- [Background] Farhad T, Sarwar MKA, Chowdhury MZ, Walid A, Sadia A, Chowdhury TK. Fast Track versus Conventional Perioperative Care Protocols in Paediatric Intestinal Stoma Closure - A Randomised Study. Afr J Paediatr Surg. 2024 Apr 1;21(2):123-128. doi: 10.4103/ajps.ajps_100_22. Epub 2023 Apr 10. PMID 38546251
- [Background] Gao R, Yang H, Li Y, Meng L, Li Y, Sun B, Zhang G, Yue M, Guo F. Enhanced recovery after surgery in pediatric gastrointestinal surgery. J Int Med Res. 2019 Oct;47(10):4815-4826. doi: 10.1177/0300060519865350. Epub 2019 Aug 4. PMID 31379230
- [Background] Al-Taher R, Alshahwan H, Abdelhadi S, Abeeleh FA, Rashdan M, Amarin M, Addasi R, Alsaraireh D, Abu-Shanab A, Alaridah N. Enhanced recovery concepts in paediatric patients who underwent appendectomy: a retrospective cohort study at a tertiary university hospital. J Int Med Res. 2023 Feb;51(2):3000605231158524. doi: 10.1177/03000605231158524. PMID 36852822